CLINICAL TRIAL: NCT02811484
Title: Efficacy of Exenatide-LAR Alone and in Combination With Dapagliflozin in Overweight/Obese, Insulin Treated Patients With Uncontrolled Type 2 Diabetes
Brief Title: Efficacy of Exenatide-LAR and Dapagliflozin in Overweight/Obese, Insulin Treated Patients With Type 2 Diabetes
Acronym: Dexlar
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to enroll due to the widespread use of both classes of drugs in patients with T2DM, including those on concomitant insulin therapy.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1512016843
Record Dates: First submitted 2016-06-17; First posted 2016-06-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Exenatide; dapagliflozin; Insulin Glargine; Insulin Detemir; Insulin Aspart; Insulin Lispro; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Other): Insulin titration and behavioral therapy.
  Interventions: Drug: Insulin Titration; Behavioral: Behavioral Therapy
- Group 2 (Placebo Comparator): Exenatide-LAR plus Dapagliflozin placebo, basal insulin titration, and behavioral therapy.
  Interventions: Drug: Exenatide-LAR plus Dapagliflozin placebo; Drug: Insulin Titration; Behavioral: Behavioral Therapy
- Group 3 (Experimental): Exenatide-LAR plus Dapagliflozin, basal insulin titration, and behavioral therapy.
  Interventions: Drug: Exenatide-LAR plus Dapagliflozin; Drug: Insulin Titration; Behavioral: Behavioral Therapy

INTERVENTIONS:
Drug: Exenatide-LAR plus Dapagliflozin placebo — Exenatide-LAR 2 mg every week x 24 weeks plus Dapagliflozin placebo x 52 weeks and behavioral therapy.
  Other Names: Bydureon; Farxiga
  Arms: Group 2
Drug: Exenatide-LAR plus Dapagliflozin — Exenatide-LAR 2 mg every week x 24 weeks plus Dapagliflozin 5 mg x 2 weeks, then 10 mg for 22 weeks and behavioral therapy.
  Other Names: Bydureon; Farxiga
  Arms: Group 3
Drug: Insulin Titration — Basal insulin titration up to 12 weeks followed by basal-bolus regimen in those with HbA1c>8%
  Other Names: Lantus, Levemir, Novolog, Lispro
Behavioral: Behavioral Therapy — Subjects will be seen by a registered dietitian and receive nutritional and lifestyle counseling according to a web-based weight management program.

SUMMARY:
The purpose of this study is to see what the effects of using one or two additional diabetes drugs (dapagliflozin and exenatide-LAR) are on blood sugar levels in patients who are taking insulin. This research study is being done to investigate which of these commonly-used medications, medication combinations or increasing insulin dose is better.

DETAILED DESCRIPTION:
This is a single center prospective, randomized, placebo-controlled trial in overweight/obese patients with insulin treated uncontrolled type 2 diabetes

Eligible subjects willing to participate in the study will be randomized to one of 3 treatment groups:

Group 1: Insulin titration + behavioral therapy Basal insulin titration upto 12 weeks with 2 U increment every 3 days (Fasting glucose goal <110) based on self-monitored blood glucose.

After 12 weeks, patients with HbA1c >8% will switch to a basal bolus regimen.

Group 2: Exenatide-LAR 2mg q week x 24 weeks + Dapagliflozin placebo x 52 weeks + titrated basal insulin +behavioral therapy.

Group 3: Exenatide-LAR 2mg q week x 24 weeks plus Dapagliflozin 5mg QD x 2 weeks followed by 10mg QD x22 weeks +titrated basal insulin + behavioral therapy.

Behavioral therapy will be delivered by registered dietitians and will include the BMIQ program -a web based medical weight loss program.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Type 2 diabetes
* BMI ≥27kg/m^2
* Hemoglobin A1C 8-12%
* English speaking
* provided written consent
* on a stable dose of metformin and/or glitazone and/or alpha-glucosidase inhibitors for ≥ to 8 weeks

Exclusion Criteria:

* History of type 1 diabetes
* fasting c-peptide <.8 ng/ml
* eGFR <60 ml/min/1.73 m^2
* urine albumin-to-creatinine ratio greater or equal to 300 mg/g
* AST/ALT greater or equal to 2.5 upper limits of normal
* history of infectious liver disease (HBV, HCV)
* creatine kinase greater or equal to 3 times the upper limits of normal
* unstable or serious cardiovascular, renal, or hepatic disease
* symptoms of severely uncontrolled diabetes
* history of more than 1 episode of severe/major hypoglycemia within 6 months, active/history of bladder cancer
* female patients who are pregnant or intending to become pregnant
* women who are breastfeeding
* personal/family history of medullary thyroid cancer or MEN2
* fasting triglyceride levels > 500 mg/dl
* history of confirmed pancreatitis
* known hypersensitivity or allergy to exenatide or dapagliflozin
* are currently enrolled in or discontinued within last 30 days from another study
* have any other condition that precludes the patient from following and completing the protocol
* history of diabetic ketoacidosis
* anti-diabetes medication other than those listed in the inclusion criteria within 8 weeks of screening
* history of previous bariatric surgery or planned bariatric surgery during the course of the study
* clinically significant abnormal free T4/TSH requiring initiation or adjustment of thyroid treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | baseline, 24 weeks
  To determine the efficacy of Exenatide-LAR and Exenatide-LAR plus dapagliflozin in lowering HbA1c compared with insulin titration in obese, insulin treated subjects with uncontrolled Type 2 Diabetes Mellitus at 24 weeks

SECONDARY OUTCOMES:
Change in Body Weight | baseline, 24 weeks
  To determine the effect of Exenatide-LAR and Exenatide-LAR plus dapagliflozin vs insulin titration on body weight in obese, insulin treated subjects with uncontrolled T2DM
Change in waist circumference | baseline, 24 weeks
  To determine the effect of Exenatide-LAR and Exenatide-LAR plus dapagliflozin vs insulin titration on waist circumference in obese, insulin treated subjects with uncontrolled T2DM
Change in fasting glucose | baseline, 24 weeks
  To determine the effect of Exenatide-LAR and Exenatide-LAR plus dapagliflozin vs insulin titration on fasting glucose (FG) in obese, insulin treated subjects with uncontrolled T2DM
Change in fasting lipids | baseline, 24 weeks
  To determine the effect of Exenatide-LAR and Exenatide-LAR plus dapagliflozin vs insulin titration on fasting lipids in obese, insulin treated subjects with uncontrolled T2DM
Change in blood pressure | baseline, 24 weeks
  To determine the effect of Exenatide-LAR and Exenatide-LAR plus dapagliflozin vs insulin titration on blood pressure in obese, insulin treated subjects with uncontrolled T2DM
Change in total dose insulin | baseline, 24 weeks
  To determine the effect of Exenatide-LAR and Exenatide-LAR plus dapagliflozin vs insulin titration on total dose insulin in obese, insulin treated subjects with uncontrolled T2DM

CONTACTS AND LOCATIONS:
Overall Officials: Alpana P Shukla, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Comprehensive Weight Control Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No